CLINICAL TRIAL: NCT01651286
Title: Determination of the Efficacy of Nasal Mask Ventilation During the Induction of General Anesthesia
Brief Title: Nasal Mask Ventilation During the Induction of General Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Yandong Jiang, Assistant Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2011P001283
Record Dates: First submitted 2012-06-06; First posted 2012-07-27 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Mechanical Ventilation Complication; Upper Airway Obstruction
Keywords: General anesthesia; Positive-pressure ventilation; Masks
MeSH Terms: conditions — Airway Obstruction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- nasal mask (Experimental): when the patient is apneic after the injection of anesthetics in the operating room, a nasal mask will be applied with positive pressure ventilation for 1 min. Then the nasal mask will be replaced with a full face mask for 1 min. Subsequently, the face mask will be replaced with the nasal mask.
  Interventions: Procedure: nasal mask; Procedure: full face mask
- full face mask (Active Comparator): when the patient is apneic after the injection of anesthetics in the operating room, a full face mask will be applied with positive pressure ventilation for 1 min. Then the full face mask will be replaced with a nasal mask for 1 min. Subsequently, the nasal mask will be replaced with the full face mask.
  Interventions: Procedure: nasal mask; Procedure: full face mask

INTERVENTIONS:
Procedure: nasal mask — Using the nasal mask instead of the full face mask during the induction of general anesthesia
Procedure: full face mask — using a standard full face mask during the induction of general anesthesia.

SUMMARY:
Recently, the investigators demonstrated that nasal route ventilation is superior to the nasal-oral combined ventilation in the absence of jaw thrust and chin up maneuvers. The investigators hypothesize nasal mask ventilation may reduce the incidence of difficult mask ventilation during the induction of general anesthesia by: 1) producing a better seal than full face mask, and 2)establishing a greater airway patency and more effectively ventilate than full face mask ventilation. The investigators intend to test this hypothesis on adult patients during the induction of general anesthesia in the absence of muscle relaxation.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age
* ASA physical status classification I-II
* general anesthesia
* elective surgery
* who are able to breathe through both their nose and mouth while awake

Exclusion Criteria:

* Patients with major cardiovascular disease, respiratory disease, cerebral vascular disease or American Society of Anesthesiologists physical status class III or greater.
* Abnormal vital signs on the day of admission for surgery [heart rate (HR, >100 bpm or <40 bpm), blood pressure (BP, >180/100 mmHg or <90/60 mmHg), room air transcutaneous oxyhemoglobin saturation (SPO2) <96%] that are not correctable with his or her routine medication or commonly used pre-operative medication.
* Unable to open mouth (<2.5 cm) or unable to breathe through their mouth or nose.
* Any person with an anticipated difficult airway. This will include subjects that require or may require either a fiberoptic intubation or intubation while awake.
* Gastric-esophageal reflex or a full stomach.
* Neurological symptoms associated with neck extension, a neurological deficit from a previous stroke or spinal cord injury, a recent stroke or Transient Ischemic Attack (TIA) within 2 weeks.
* Pregnant women and women less than one month post-partum. Ruling out pregnancy will be conducted by careful history and physical examination as performed routinely prior to surgery. If the history is believed to be unreliable, the patient will be excluded unless a pregnancy test is performed and the result of the test is negative.
* Emergency cases and subjects who have not adhered to the ASA NPO (Nil Per Os - Nothing By Mouth) guidelines.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2012-06; Primary Completion 2013-06 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Tidal volume | in 30 minutes after the induction of general anesthesia
  Tidal volume generated by the positive pressure ventilation during the induction of general anesthesia

SECONDARY OUTCOMES:
Carbon dioxide removal | in 30 minutes after the induction of general anesthesia
  carbon dioxide removed per minute during the induction of general anesthesia will be calculated
success rate of positive pressure ventilation with different masks | in 30 minute after the induction of general anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Hovig V Chitilian, MD, Principal Investigator — Massachusetts General Hospital; Yandong Jiang, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States